CLINICAL TRIAL: NCT02906735
Title: Evaluation of Static and Dynamic Foot Pressure Measurement After Implantation of Knee Joint Prostheses or Alignment Surgeries of the Knee
Brief Title: Changes of Plantar Pressure After Knee Reconstructive Surgery
Acronym: PEDKnee
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Harrasser, Principal Investigator, Technical University of Munich
Other Study IDs: TUM1
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-09

CONDITIONS: Knee Pain Treated With Knee Arthroplasty
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Patients with knee surgery undergo plantar foot pressure measurement pre- and postoperatively
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Implantation of knee joint prosthesis or deviation osteotomies of the knee

SUMMARY:
Knee reconstructive surgery (knee prosthesis, osteotomies) often results in changes of alignment of the lower limb axis. This affects also biomechanics of the hindfoot. There is a lack of understanding what changes of alignment of the lower limb causes to the ankle. The investigators want to evaluate the effects of knee surgeries onto the plantar foot pressure investigated by means of static and dynamic pedography.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for knee surgery willing to participate at this study

Exclusion Criteria:

* No informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients planned for knee surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Foot pressure curve preoperatively | -1 day
  scale

SECONDARY OUTCOMES:
Foot pressure curve postoperatively | 1 year
  scale

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Harrasser, Principal Investigator — Klinikum rechts der Isar
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided